CLINICAL TRIAL: NCT01746485
Title: A PK Evaluation of Three Times Daily Dosing of UT-15C SR Tablets in Healthy Subjects
Brief Title: Three Times Daily Dosing of UT-15C
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: TDE-DU-102
Record Dates: First submitted 2012-08-16; First posted 2012-12-11 (Estimated); Last update posted 2012-12-12 (Estimated); Status verified 2012-12

CONDITIONS: Healthy
Keywords: Volunteers
MeSH Terms: interventions — treprostinil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- UT-15C (Experimental)
  Interventions: Drug: UT-15C

INTERVENTIONS:
Drug: UT-15C
  Other Names: treprostinil diethanolamine; treprostinil diolamine; UT-15C SR

SUMMARY:
To evaluate the pharmacokinetics of three-times daily dosing of UT-15C in healthy volunteers

ELIGIBILITY:
* Healthy male and female subjects
* aged 18-55 years of age;
* weight between 50 and 100 kg, with a body mass index (BMI) between 19.0 and 29.9 kg/m2, inclusive for female subjects and
* weight between 50 and 120 kg, with a BMI between 19.0 and 32.0 kg/m², inclusive for male subjects.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2012-07; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) from 0-24hrs after 6 days of TID dosing. | 6 days
  Cmax, tmax, AUC(0-6), AUC(0-24), AUC(6-12), AUC(12-24) and t1/2

SECONDARY OUTCOMES:
PK profile of UT-15C after a single 0.5mg dose on Day 1 | 1 day
  Day 1: Cmax, tmax, AUC(0-6), AUC(0-24), AUC(0-t), AUC(0-inf), and t1/2

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Pham, MD, Principal Investigator — PPD Development, LP
Locations (1):
- PPD Development, Austin, Texas, United States

REFERENCES:
- [Derived] Jones A, Wang-Smith L, Pham T, Laliberte K. Pharmacokinetics of 3 times a day dosing of oral treprostinil in healthy volunteers. J Cardiovasc Pharmacol. 2014 Mar;63(3):227-32. doi: 10.1097/FJC.0000000000000039. PMID 24603117